CLINICAL TRIAL: NCT04934722
Title: A Phase 3, Randomized, Double-blind Trial of Pembrolizumab (MK-3475) Plus Enzalutamide Plus ADT Versus Placebo Plus Enzalutamide Plus ADT in Participants With Metastatic Hormone-Sensitive Prostate Cancer (mHSPC) (KEYNOTE-991)
Brief Title: Efficacy and Safety of Pembrolizumab (MK-3475) Plus Enzalutamide Plus Androgen Deprivation Therapy (ADT) Versus Placebo Plus Enzalutamide Plus ADT in Participants With Metastatic Hormone-Sensitive Prostate Cancer (mHSPC) (MK-3475-991/KEYNOTE-991)-China Extension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3475-991 China Extension; MK-3475-991 China Extension (Other: MSD); KEYNOTE-991 (Other: MSD); jRCT2080225171 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-06-17; First posted 2021-06-22 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Hormone-Sensitive Prostate Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1),; Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; enzalutamide; Androgen Antagonists

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pembrolizumab + Enzalutamide + ADT (Experimental): Starting on Day 1 of each 21-day cycle, participants receive 200 mg pembrolizumab intravenously (IV) every 3 weeks (Q3W) for up to 35 cycles (approximately 2 years), plus 160 mg enzalutamide taken orally once daily, while maintaining continuous ADT with a luteinizing-hormone releasing hormone (LHRH) agonist or antagonist during study treatment. Participants will continue to receive enzalutamide and ADT until criteria for discontinuation are met.
  Interventions: Biological: Pembrolizumab; Drug: Enzalutamide; Drug: Androgen Deprivation Therapy (ADT)
- Placebo + Enzalutamide + ADT (Placebo Comparator): Starting on Day 1 of each 21-day cycle, participants receive placebo IV Q3W for up to 35 cycles (approximately 2 years), plus 160 mg enzalutamide taken orally once daily, while maintaining continuous ADT with a LHRH agonist or antagonist during study treatment. Participants will continue to receive enzalutamide and ADT until criteria for discontinuation are met.
  Interventions: Drug: Enzalutamide; Drug: Androgen Deprivation Therapy (ADT); Other: Placebo

INTERVENTIONS:
Biological: Pembrolizumab — Pembrolizumab is administered as an IV infusion at 200 mg on Day 1 of each 21-day cycle for up to 35 cycles.
  Other Names: KEYTRUDA®; MK-3475
  Arms: Pembrolizumab + Enzalutamide + ADT
Drug: Enzalutamide — Enzalutamide is administered orally as capsules/tablets at a dosage of 160 mg daily. Enzalutamide is administered continuously until criteria for discontinuation are met.
  Other Names: XTANDI®
Drug: Androgen Deprivation Therapy (ADT) — Stable regimen of ADT (LHRH agonist or antagonist) at a dose and frequency of administration that is consistent with the local product label.
Other: Placebo — Placebo infusion solution is administered as an IV infusion on Day 1 of each 21-day cycle for up to 35 cycles.
  Arms: Placebo + Enzalutamide + ADT

SUMMARY:
This study will assess the efficacy and safety of pembrolizumab plus enzalutamide plus ADT versus placebo plus enzalutamide plus ADT in Chinese participants with mHSPC. The primary hypothesis is that in participants with mHSPC, the combination of pembrolizumab plus enzalutamide plus ADT is superior to placebo plus enzalutamide plus ADT with respect to 1) radiographic progression-free survival (rPFS) per Prostate Cancer Working Group (PCWG)-modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as assessed by blinded independent central review (BICR) and 2) overall survival (OS). As of Amendment 4, the study is being stopped for futility. All the prespecified interim analysis after interim analysis (IA1) and final analysis of the study described the statistical analysis plan (SAP) will not be performed. Safety analysis will be performed at the end of the study; there will be no further analyses for efficacy and electronic patient-reported outcome (ePRO) endpoints collected from participants beyond the IA1 cutoff date. All study participants will stop ongoing treatment with pembrolizumab/placebo. Exceptions may be requested for study participants who, in the assessment of their study physician, are benefitting from the combination of enzalutamide and pembrolizumab, after consulting with the Sponsor. All other study participants should be discontinued from study and be offered standard of care (SOC) treatment as deemed necessary by the Investigator. If enzalutamide as SOC is not accessible off study to the participant, central sourcing may continue. As of Amendment 04, disease progression will no longer be centrally verified, participants will only be assessed locally. As of Amendment 4, Second Course treatment is not an option for participants. There are currently no participants in the Second Course Phase.

DETAILED DESCRIPTION:
The China extension study will include participants previously enrolled in China in the global study for MK-3475-991 (NCT04191096) plus those enrolled during the China extension enrollment period. A total of approximately 186 Chinese participants will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Male participants with histologically- or cytologically-confirmed adenocarcinoma of the prostate without small cell histology
* Has metastatic disease assessed by investigator and verified by BICR by either ≥2 bone lesions on bone scan and/or visceral disease by computed tomography/magnetic resonance imaging (CT/MRI)
* Willing to maintain continuous Androgen Deprivation Therapy (ADT) with a luteinizing-hormone releasing hormone (LHRH) agonists or antagonists during study treatment or have a history of bilateral orchiectomy
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 assessed within 10 days of randomization
* Participants receiving bone resorptive therapy (including, but not limited to, bisphosphonate or denosumab) must have been on stable doses prior to randomization
* Has adequate organ function
* Has provided newly obtained core or excisional biopsy (obtained within 12 months of screening) from soft tissue not previously irradiated (samples from tumors progressing in a prior site of radiation are allowed). Participants with bone only or bone predominant disease may provide a bone biopsy sample
* Male participants must agree to the following during the intervention period and for at least 120 days after the last dose of study intervention: Refrain from donating sperm PLUS either be abstinent from heterosexual intercourse and agree to remain abstinent OR agree to use contraception, unless confirmed to be azoospermic
* Male participants must agree to use male condom when engaging in any activity that allows for passage of ejaculate to another person of any sex

Exclusion Criteria:

* Has a known additional malignancy that is progressing or has required active treatment in the last 3 years
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy
* Has undergone major surgery including local prostate intervention (excluding prostate biopsy) within 28 days prior to randomization and not recovered adequately from the toxicities and/or complications
* Has a gastrointestinal disorder affecting absorption or is unable to swallow tablets/capsules
* Has an active infection (including tuberculosis) requiring systemic therapy
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has known active human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Has known or suspected central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has a history of seizure or any condition that may predispose to seizure
* Has a history of loss of consciousness within 12 months of screening
* Has had myocardial infarction or uncontrolled angina within 6 months prior to randomization, or has New York Heart Association class III or IV congestive heart failure or a history of New York Heart Association class III or IV congestive heart failure
* Has hypotension (systolic blood pressure <86 millimeters of mercury [mmHg]) or uncontrolled hypertension (systolic blood pressure >170 mmHg or diastolic blood pressure >105 mmHg) at the screening visit
* Has a history of clinically significant ventricular arrhythmias
* Has hypersensitivity to pembrolizumab and/or enzalutamide and/or any of their excipients
* Has received prior ADT as neoadjuvant/adjuvant therapy for non-metastatic prostate cancer for >39 months in duration or within 9 months prior to randomization or with evidence of disease progression while receiving ADT
* Has had prior treatment with a next generation hormonal agent (eg, abiraterone, enzalutamide, apalutamide, darolutamide)
* Has received prior therapy with an anti-programmed cell death-1 (anti-PD-1), anti-programmed cell death-ligand 1 (anti-PD-L1), or anti-programmed cell death-ligand 2 (anti PD-L2) agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor
* Has received a live vaccine within 30 days prior to randomization
* Has a "superscan" bone scan
* Has had an allogenic tissue/solid organ transplant
* Is expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment
* Has received any prior pharmacotherapy, radiation therapy or surgery for metastatic prostate cancer with the following exceptions:

  1. Up to 3 months of ADT or orchiectomy with or without concurrent first-generation antiandrogens, if patient was not treated with docetaxel
  2. May have 1 course of palliative radiation or surgical therapy to treat symptoms resulting from metastatic disease if it was administered at least 4 weeks prior to randomization
  3. For participants with low volume metastatic disease, may have 1 course of definitive radiotherapy if it was administered at least 4 weeks prior to randomization
  4. Up to 6 cycles of docetaxel therapy with final treatment administration completed within 2 months of randomization and no evidence of disease progression. In these participants up to 6 months of ADT permitted

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2025-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (24):
- China (24):
  - Peking University First Hospital ( Site 0800), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 0802), Beijing, Beijing Municipality
  - Chongqing Cancer Hospital ( Site 0815), Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University (Site 0816), Xiamen, Fujian
  - Sun Yat-Sen University Cancer Center ( Site 0825), Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University-Urology ( Site 0638), Guangzhou, Guangdong
  - Sun Yat Sen Memorial Hospital (Site # 0819), Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital ( Site 0838), Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital ( Site 0822), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 0818), Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology ( Site 0829), Wuhan, Hubei
  - Hubei Cancer Hospital ( Site 0833), Wuhan, Hubei
  - Hunan Cancer Hospital ( Site 0817), Changsha, Hunan
  - Nanjing Drum Tower Hospital ( Site 0811), Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University ( Site 0821), Nanchang, Jiangxi
  - The Second Affiliated Hosp of Xi'an Jiaotong Univ College of Medicine ( Site 0831), Xi'an, Shaanxi
  - Renji Hospital Shanghai Jiaotong University School of Medicine ( Site 0807 ), Shanghai, Shanghai Municipality
  - The first affiliated Hospital of Xi an Jiaotong University ( Site # 0812), Xi’an, Shanxi
  - Tianjin Medical University Cancer Institute & Hospital ( Site 0804 ), Tianjin, Tianjin Municipality
  - 2nd Affil Hosp of Zhejiang University College of Medicine ( Site 0808), Hangzhou, Zhejiang
  - The 1st Affil Hosp of College of Medicine, Zhejiang Univ ( Site 0830), Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital ( Site 0809), Hangzhou, Zhejiang
  - Ningbo First Hospital-Urology (0835), Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University ( Site 0834), Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 186 Chinese participants were randomized and received treatment (global study [NCT04191096; n =7] and to the extension portion [n=179]). All safety results were reported on all participants treated.
Groups:
- Pembrolizumab + Enzalutamide + ADT: Participants received 200 mg pembrolizumab IV on Day 1 of each 3-week cycle for up to 35 cycles (approximately 2 years), plus 160 mg enzalutamide taken orally once daily (QD), while maintaining continuous ADT with a luteinizing-hormone releasing hormone (LHRH) agonist or antagonist during study treatment. Participants received enzalutamide and ADT until criteria for discontinuation were met.
- Placebo + Enzalutamide + ADT: Participants received placebo IV on Day 1 of each 3-week cycle for up to 35 cycles (approximately 2 years), plus 160 mg enzalutamide taken orally QD, while maintaining continuous ADT with a LHRH agonist or antagonist during study treatment. Participants received enzalutamide and ADT until criteria for discontinuation are met
Period: Overall Study
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Started | 92 | 94
Completed | 0 | 0
Not Completed | 92 | 94
Not completed — Death | 4 | 3
Not completed — Participants Ongoing | 88 | 91

BASELINE CHARACTERISTICS:
Population: All Chinese participants who were randomized to the global study (NCT04191096) and to the extension portion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT | Total
Number analyzed (Participants) | 92 | 94 | 186
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.5 (7.1) | 67.4 (7.6) | 67.9 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 92 | 94 | 186
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 92 | 94 | 186
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 92 | 94 | 186
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Progression-free Survival (rPFS) Per Prostate Cancer Working Group (PCWG)-Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: rPFS was defined as the time from randomization to occurrence of: radiological tumor progression using RECIST 1.1 as assessed by BICR; progression of bone lesions using PCWG criteria; or death due to any cause. Progression as per modified RECIST 1.1 was ≥20% increase in sum of diameters of target lesions and progression of existing non-target lesions. Progression of bone lesions by PCWG criteria was the appearance of ≥2 new bone lesions on bone scan, that have been confirmed to not represent tumor flare, and was persistent for ≥6 weeks. The rPFS was calculated using the product-limit (Kaplan-Meier) method for censored data. Participants without a rPFS event were censored at the date of last disease assessment.
Time Frame: Up to approximately 17 months
Population: All Chinese participants who were randomized to the global study (NCT04191096) or to the extension portion that were evaluable for response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 92 | 94
Months | 14.4 [NA to NA] — NA = lower limit and upper limit of 95% CI for rPFS cannot be calculated at the time of last disease assessment due to insufficient number of participants with events. | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for rPFS cannot be calculated at the time of last disease assessment due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide + ADT vs Placebo + Enzalutamide + ADT; Test type: Other; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.24 to 2.34] — HR and associated 95% Confidence Interval (CI) were calculated using Cox regression model with Efron's method of tie handling with treatment as a covariate

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. The OS was calculated using the product-limit (Kaplan-Meier) method for censored data. Participants without documented death at the time of the analysis were censored at the date of the last follow-up.
Time Frame: Up to approximately 17 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 92 | 94
Months | NA [14.4 to NA] — NA = Median and upper limit of 95% CI for OS cannot be calculated at the time of last disease assessment due to insufficient number of participants with events. | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for OS cannot be calculated at the time of last disease assessment due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide + ADT vs Placebo + Enzalutamide + ADT; Test type: Other; Hazard Ratio (HR) = 1.35, 95% CI 2-sided [0.30 to 6.01] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Time to Initiation of the First Subsequent Anti-cancer Therapy or Death (TFST)
Description: TFST was defined as the time from randomization to initiation of the first subsequent anti-cancer therapy or death; whichever occurred first. The TFST was calculated using the product limit (Kaplan-Meier) method for censored data. Participants without documented event at time of analysis will be censored at the date of last known time to have not received subsequent new anti-cancer therapy.
Time Frame: Up to Approximately 17 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 92 | 94
Months | NA [14.4 to NA] — NA = Median and upper limit of 95% CI for TFST cannot be calculated at the time of last disease assessment due to insufficient number of participants with events | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for TFST cannot be calculated at the time of last disease assessment due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide + ADT vs Placebo + Enzalutamide + ADT; Test type: Other; Hazard Ratio (HR) = 1.35, 95% CI 2-sided [0.50 to 3.63] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Time to First Symptomatic Skeletal-related Event (TTSSRE)
Description: TTSSRE was the time from randomization to the first symptomatic skeletal-related event defined as: use of external-beam radiation therapy (EBRT) to prevent or relieve skeletal symptoms, occurrence of new symptomatic pathologic bone fracture (vertebral or nonvertebral), occurrence of spinal cord compression, or tumor-related orthopedic surgical intervention, whichever occurs first. The TTSSRE was calculated using the Kaplan-Meier method for censored data. Participants without symptomatic skeletal-related events were censored at the last evaluable assessment.
Time Frame: Up to Approximately 17 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 92 | 94
Months | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for TTSSRE cannot be calculated at the time of last disease assessment due to insufficient number of participants with events. | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for TTSSRE cannot be calculated at the time of last disease assessment due to insufficient number of participants with events.

5. Secondary Outcome: Time to Prostate-specific Antigen (PSA) Progression
Description: Time to PSA progression was the time from randomization to PSA progression. The PSA progression date was defined as the date of 1) ≥25% increase and ≥2 ng/mL above the nadir, confirmed by a second value ≥3 weeks later if there is PSA decline from baseline, or 2) ≥25% increase and ≥2 ng/mL increase from baseline beyond 12 weeks if there is no PSA decline from baseline. Time to PSA was calculated using Kaplan-Meier method for censored data. Participants without PSA progression were censored at the last PSA date.
Time Frame: Up to Approximately 17 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 92 | 94
Months | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for Time to PSA Progression cannot be calculated at the time of last disease assessment due to insufficient number of participants with events | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for Time to PSA Progression cannot be calculated at the time of last disease assessment due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide + ADT vs Placebo + Enzalutamide + ADT; Test type: Other; Hazard Ratio (HR) = 3.15, 95% CI 2-sided [0.33 to 30.29] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Time to Radiographic Soft Tissue Progression Per Soft Tissue Rules of PCWG-Modified RECIST 1.1 as Assessed by BICR
Description: The time to radiographic soft tissue progression was defined as the time from randomization to radiographic soft tissue progression per soft tissue rules of PCWG-modified RECIST 1.1 as assessed by BICR. Progression was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered progression. Time to radiographic soft tissue progression was calculated using the product-limit (Kaplan-Meier) method for censored data. Participants without radiographic soft tissue progression were censored at the last evaluable assessment.
Time Frame: Up to Approximately 17 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 92 | 94
Months | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for time to radiographic soft tissue progression cannot be calculated at the time of last disease assessment due to insufficient number of participants with events | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for time to radiographic soft tissue progression cannot be calculated at the time of last disease assessment due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide + ADT vs Placebo + Enzalutamide + ADT; Test type: Other; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.11 to 4.07] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Time to Pain Progression (TTPP) as Assessed by Brief Pain Inventory-Short Form (BPI-SF) Item #3 ("Worst Pain in 24 Hours") and Opiate Use
Description: TTPP was defined as the time from randomization to pain progression as determined by Item 3 of the BPI-SF. Pain progression was defined as: 1) For participants asymptomatic at baseline: a >2-point change from baseline in the average BPI-SF item 3 score at 2 consecutive visits or initiation of opioid use for pain 2) For participants symptomatic at baseline (average BPI-SF Item 3 score >0 and/or currently taking opioids; a >2-point change from baseline in the average BPI-SF Item 3 score and the average worst pain score >4 and no decrease in average opioid use. TTPP was calculated using the Kaplan-Meier method for censored data. Participants who had > 2 consecutive visits that were not evaluable for pain progression were censored at the last evaluable assessment.
Time Frame: Up to Approximately 17 months
Population: All Chinese participants who were randomized to the global study (NCT04191096) or to the extension portion who received at least one dose of study treatment, and who had at least 1 BPI-SF assessment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 91 | 91
Months | NA [9.4 to NA] — NA = Median and upper limit of 95% CI for TTPP cannot be calculated at the time of last disease assessment due to insufficient number of participants with events | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for TTPP cannot be calculated at the time of last disease assessment due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide + ADT vs Placebo + Enzalutamide + ADT; Test type: Other; Hazard Ratio (HR) = 1.45, 95% CI 2-sided [0.73 to 2.90] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Time From Randomization to Disease Progression as Determined by Investigator Assessment After Next-line of Therapy or Death From Any Cause, Whichever Occurs First (PFS2)
Description: PFS2 was defined as the time from randomization to disease progression as determined by investigator assessment of radiological or clinical progression after next-line of therapy or death from any cause, whichever occurs first.
Time Frame: Up to Approximately 17 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 92 | 94
Months | NA [14.4 to NA] — NA = Median and upper limit of 95% CI for PFS2 cannot be calculated at the time of last disease assessment due to insufficient number of participants with events | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for PFS2 cannot be calculated at the time of last disease assessment due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide + ADT vs Placebo + Enzalutamide + ADT; Test type: Other; Hazard Ratio (HR) = 1.75, 95% CI 2-sided [0.42 to 7.34] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Prostate-specific Antigen (PSA) Response Rate
Description: PSA response rate was the percentage of participants who had PSA response defined as a reduction in the PSA level from baseline by >50%. The reduction in PSA level was confirmed by an additional PSA evaluation performed >3 weeks from the original response.
Time Frame: Up to Approximately 17 Months
Population: All Chinese participants who were randomized to the global study (NCT04191096) or to the extension portion who had a baseline PSA measurement and had data available for analysis
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 92 | 94
Percentage of Participants | 93.5 [86.3 to 97.6] | 98.9 [94.2 to 100.0]
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide + ADT vs Placebo + Enzalutamide + ADT; Test type: Other; Percent Difference = -5.5, 95% CI 2-sided [-12.6 to 0.0] — Percent difference and associated 95% CI were calculated using Miettinen & Nurminen method

10. Secondary Outcome: Prostate-specific Antigen (PSA) Undetectable
Description: PSA undetectable rate was defined as the percentage of participants with detectable PSA (> 0.2 ng/mL) at baseline, which becomes undetectable (< 0.2 ng/mL) during study treatment.
Time Frame: Up to Approximately 17 Months
Population: All Chinese participants who were randomized to the global study (NCT04191096) or to the extension portion with detectable PSA at baseline and had data available for analysis
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 90 | 93
Percentage of Participants | 45.6 [35.0 to 56.4] | 46.2 [35.8 to 56.9]
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide + ADT vs Placebo + Enzalutamide + ADT; Test type: Other; Percent difference = -0.7, 95% CI 2-sided [-15.0 to 13.7] — Percent difference and associated 95% CI were calculated using Miettinen & Nurminen method

11. Secondary Outcome: Objective Response Rate (ORR) Per PCWG-Modified RECIST 1.1 as Assessed by BICR
Description: ORR was defined as the percentage of participants with complete response (CR: disappearance of all target lesions per RECIST 1.1; and no evidence of disease (NED) on base scan per PCWG) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions per RECIST 1.1; and non-progressive disease, non-evaluable [NE], or NED on bone scan or CR with non-progressive disease or NE bone scan per PCWG).
Time Frame: Up to Approximately 17 Months
Population: All Chinese participants who were randomized to the global study (NCT04191096) or to the extension portion with measurable disease at baseline and had data available for analysis
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 38 | 44
Percentage of Participants | 73.7 [56.9 to 86.6] | 65.9 [50.1 to 79.5]
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide + ADT vs Placebo + Enzalutamide + ADT; Test type: Other; Percent difference = 7.8, 95% CI 2-sided [-12.5 to 27.1] — Percent difference and associated 95% CI were calculated using Miettinen & Nurminen method

12. Secondary Outcome: Duration of Response (DOR) Per PCWG- Modified RECIST 1.1 as Assessed by BICR
Description: DOR was defined as the time from first documented evidence of complete response (CR) or partial response (PR) per PCWG and RECIST 1.1 criteria until progressive disease (PD) or death. PD per RECIST 1.1 was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of a least 5 mm. PD per PCWG was the appearance of >2 new bone lesions on bone scan, that have been confirmed to not represent tumor flare, and were persistent for >6 weeks. The DOR was calculated using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to Approximately 17 Months
Population: All Chinese participants who were randomized to the global study (NCT04191096) or to the extension portion who demonstrated a CR or PR, and had data available for analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 38 | 44
Months | NA [5.8 to NA] — NA = Median and upper limit of 95% CI for DOR cannot be calculated at the time of last disease assessment due to insufficient number of participants with response | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for DOR cannot be calculated at the time of last disease assessment due to insufficient number of participants with response

13. Secondary Outcome: Number of Participants Who Experience an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could therefore have been any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. Participants who experienced an AE will be reported for each arm.
Time Frame: Up to Approximately 17 Months
Reporting Status: Not Posted, anticipated posting 2027-06

14. Secondary Outcome: Number of Participants Who Discontinue Study Treatment Due to an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinue study treatment due to an AE will be reported for each arm.
Time Frame: Up to Approximately 17 Months
Reporting Status: Not Posted, anticipated posting 2027-06

ADVERSE EVENTS:
Time Frame: Up to approximately 17 months
Description: All-cause mortality was reported on all randomized participants and adverse events (serious and non-serious) were reported on all participants who received ≥1 dose of treatment. Per protocol, disease progression was not considered an AE unless related to treatment. Medical Dictionary for Regulatory Activities (MedDRA) terms neoplasm progression, malignant neoplasm progression, and disease progression not related to treatment were excluded.
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
All-Cause Mortality (participants affected / at risk) | 4/92 | 3/94
Serious Adverse Events (participants affected / at risk) | 24/92 | 10/94
Other Adverse Events (participants affected / at risk) | 79/92 | 79/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Enzalutamide + ADT (N=92) | Placebo + Enzalutamide + ADT (N=94)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Autoimmune myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0)
Immune-mediated thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (3) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Immune-mediated nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Enzalutamide + ADT (N=92) | Placebo + Enzalutamide + ADT (N=94)
Anaemia (Blood and lymphatic system disorders) | 25 (34) | 14 (19)
Hypothyroidism (Endocrine disorders) | 9 (9) | 4 (6)
Constipation (Gastrointestinal disorders) | 7 (7) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 8 (10) | 7 (8)
Nausea (Gastrointestinal disorders) | 4 (4) | 7 (7)
Toothache (Gastrointestinal disorders) | 3 (4) | 6 (6)
Fatigue (General disorders) | 9 (9) | 7 (8)
Malaise (General disorders) | 10 (10) | 4 (5)
Pyrexia (General disorders) | 8 (8) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 8 (8)
Alanine aminotransferase increased (Investigations) | 18 (20) | 21 (22)
Aspartate aminotransferase increased (Investigations) | 14 (16) | 17 (17)
Blood alkaline phosphatase increased (Investigations) | 5 (5) | 5 (6)
Blood bilirubin increased (Investigations) | 4 (5) | 5 (9)
Blood cholesterol increased (Investigations) | 6 (7) | 2 (2)
Blood thyroid stimulating hormone increased (Investigations) | 5 (6) | 8 (10)
Lymphocyte count decreased (Investigations) | 2 (2) | 5 (6)
Neutrophil count decreased (Investigations) | 5 (9) | 1 (8)
Platelet count decreased (Investigations) | 10 (19) | 10 (17)
Weight decreased (Investigations) | 4 (4) | 5 (5)
Weight increased (Investigations) | 8 (8) | 12 (15)
White blood cell count decreased (Investigations) | 7 (12) | 5 (10)
Decreased appetite (Metabolism and nutrition disorders) | 11 (11) | 5 (5)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 (7) | 4 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 16 (26) | 20 (33)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (5) | 6 (8)
Hyperlipidaemia (Metabolism and nutrition disorders) | 8 (13) | 7 (9)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6 (8) | 4 (5)
Hyperuricaemia (Metabolism and nutrition disorders) | 5 (8) | 6 (7)
Hypocalcaemia (Metabolism and nutrition disorders) | 7 (8) | 6 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (10) | 6 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (9) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (10) | 11 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 9 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (9) | 8 (9)
Dizziness (Nervous system disorders) | 9 (11) | 7 (7)
Headache (Nervous system disorders) | 5 (7) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 5 (7) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (3)
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 7 (8) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 23 (29) | 9 (10)
Hot flush (Vascular disorders) | 8 (8) | 9 (9)
Hypertension (Vascular disorders) | 14 (16) | 11 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor will comply with the requirements for publication of study results. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT04934722/Prot_SAP_000.pdf